CLINICAL TRIAL: NCT01653054
Title: The Incidence of Abnormal Anal Pap Smears in Patients With Inflammatory Bowel Disease
Brief Title: Anal Dysplasia in Patients With Inflammatory Bowel Disease
Acronym: HPVIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-01-050E
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: IBD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBD patients ON Immunosuppression (Experimental)
  Interventions: Procedure: Anal Pap Smear, HPV DNA Testing
- IBD Patients OFF Immunosuppression (Experimental)
  Interventions: Procedure: Anal Pap Smear, HPV DNA Testing

INTERVENTIONS:
Procedure: Anal Pap Smear, HPV DNA Testing — Anal Pap Smears and HPV DNA testing will be performed on all subjects.

SUMMARY:
The rationale for this study is that the risk of anal dysplasia in patients with inflammatory bowel disease (IBD) as compared to the general population has yet to be investigated prospectively. There have only been a few articles examining this relationship - preliminary results have suggested that patients with IBD are at increased risk for abnormal anal pap smears. As high grade anal dysplasia is strongly associated with an increased risk of anal carcinoma, it is important to identify all high risk groups that might benefit from routine screening. This pilot study aims to determine whether patients with IBD in our Bronx population have an increased risk of abnormal anal Pap smears. We hypothesize that there will be an increased incidence of abnormal anal pap smears in patients with IBD who have been treated with immunosuppressants, given that chronic immunosuppression is related to increased HPV infection.

DETAILED DESCRIPTION:
IBD patients on and off immunosuppression will be identified from gastroenterology fellow clinics. After patients express interest in the study, a study coordinator will provide an overview of the study and obtain consent prior to initiating any research related procedures. Anal Pap smears and Digene Hybrid Capture 2 High-Risk HPV DNA Tests will be performed on each study patient.

Medications will be documented for all IBD subjects and controls. Patient characteristics that will be documented will include IBD diagnosis, area of involvement (small bowel vs. large bowel, rectal involvement), type and duration of immunosuppressant use, smoking status, family history of any dysplasia (including anus), and reproductive risk factors. Data will be reported by subjects in subject interviews and through questionnaires.

For the purposes of analysis, subjects will be divided into two groups: IBD patients on immunosuppression and IBD patients not on immunosuppression. Results will be recorded in relation to exposure to immunosuppressive agents including prednisone, purine analogs (azathioprine/6MP), methotrexate, and infliximab. Immunosuppression will be defined as a history of at least three months of azathioprine/6MP, eight consecutive weeks of prednisone greater than 15mg per day, a cumulative dose of greater than 100mg of methotrexate, or at least one infusion of infliximab within 8 weeks of the date of the anal Pap smear. Since this is a pilot project, we will recruit a minimum of 20 subjects to each group.

Abnormalities will be classified in standard Bethesda classifications as atypical squamous cells of undetermined significance (ASCUS), low grade squamous intraepithelial lesion (LSIL), high grade squamous intraepithelial lesion (HSIL) or carcinoma. The pathologist reading the Pap smears will be blinded to the patient status (IBD versus control) and immunomodulator history.

ELIGIBILITY:
Inclusion Criteria:

* i. Women and men between the ages of 18-65 with a history of inflammatory bowel disease confirmed histologically and on immunosuppression defined as at least three months of azathioprine/6MP, eight consecutive weeks of prednisone greater than 15mg per day, a cumulative dose of greater than 100mg of methotrexate, or at least one infusion of infliximab within 8 weeks of the date of the anal Pap smear.

ii. Women and men between the ages of 18-65 with a history of inflammatory bowel disease confirmed histologically and not on immunosuppression (defined as above)

Exclusion Criteria:

* i. Patients with HIV, transplant recipients, men who have sex with men as they already represent high risk groups ii. Women with a history of an abnormal cervical Pap test within the past 2 years.

iii. Patients with active proctitis as defined by an abnormal sigmoidoscopy or colonoscopy, rectal bleeding or tenesmus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Abnormal anal cytology and presence of high risk HPV DNA | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Brandt, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York